CLINICAL TRIAL: NCT00159367
Title: The Use of Repetitive Magnetic Stimulation for Strength Training of the Quadriceps Muscle in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: The Use of Repetitive Magnetic Stimulation for Strength Training of the Quadriceps Muscle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Magstim Company, Whitland, Wales (Unknown)
Responsible Party: Professor Michael I Polkey, Royal brompton Hospital/Imperial College
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RR1; EU QLRT-2001-2285
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Neuromuscular electrical stimulation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

INTERVENTIONS:
Device: Repetitive magnetic stimulation to the quadriceps

SUMMARY:
We intend to use repetitive magnetic stimulation to the quadriceps muscle to try to improve strength and improve the metabolic function of the muscle.

DETAILED DESCRIPTION:
Quadriceps strength is reduced in COPD. Increasing quadriceps strength is one of the goals of pulmonary rehabilitation yet some patients with severe COPD are unable to exercise with sufficient intensity, due to breathlessness, to achieve a true training benefit.

Transcutaneous electrical stimulation of the femoral nerve has been shown to improve quadriceps muscle strength, muscle mass, and performance in patients with severe COPD. Magnetic stimulation may be preferred because it offers the opportunity to train the whole muscle and because it is painless. In this pilot study we are investigating whether repetitive magnetic stimulation camn increase the strength of the quadriceps muscle and whether it confers any change in structure or metabolism of the muscle itself.

ELIGIBILITY:
Inclusion Criteria:

Chronic Obstructive Pulmonary Disease

Exclusion Criteria:

Aspirin therapy Cardiac Pacemaker

-

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2005-01; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Quadriceps Twitch force

SECONDARY OUTCOMES:
Quadriceps maximal voluntary contraction, Oxidative enzyme profile, fibre type distribution and capillarity of the muscle, quality of life questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Michael I Polkey, PhD, Principal Investigator — Imperial College London
Locations (1):
- Royal Brompton Hospital, London, United Kingdom